CLINICAL TRIAL: NCT03392844
Title: Beds for Kids Program: Impact on Child Sleep and Family Functioning in Young Children
Brief Title: Impact of Beds for Kids Program on Child Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-014350
Record Dates: First submitted 2017-12-24; First posted 2018-01-08 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Insufficient Sleep Syndrome; Inadequate Sleep Hygiene; Child Behavior Problems; Emotional Stress
MeSH Terms: conditions — Sleep Deprivation; Stress, Psychological | interventions — Beds

STUDY DESIGN:
Intervention Model Description: Caregiver-child dyads will be assigned to the intervention group, in which they receive a bed through the Beds for Kids program after a 7-day period, or to the waitlist control group, in which they receive a bed after a 14-day period.
Who Masked: Outcomes Assessor
Masking Description: Research team members who are responsible for the assessment of study outcomes will be blinded to group condition. Blinding of the Lead Investigator is not possible due to the need to coordinate intervention with the Beds for Kids program. Blinds of the participants is not possible due to the nature of the intervention (scheduling and provision of beds).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Bed after 7 days (Experimental): Caregiver-child dyads in this condition will receive a bed, bedding, and sleep education from the Beds for Kids program 7 days after initiating daily diary/actigraph procedures.
  Interventions: Other: Beds for Kids program
- Wait-list: Bed after 14 days (Experimental): Caregiver-child dyads in this condition will receive a bed, bedding, and sleep education from the Beds for Kids program 14 days after initiating daily diary/actigraph procedures.
  Interventions: Other: Beds for Kids program

INTERVENTIONS:
Other: Beds for Kids program — The Beds for Kids program, which is part of the non-profit organization One House at a Time, gives every child in the program a new twin-size bed mattress, metal bed frame, and a "bedtime bag," which contains a sheet set, blanket, pillow, several books, stuffed animal, and toothbrush. Children also receive educational messages about healthy sleep habits via a magnet and "color-your-own" bookmark. All of the items are sorted, packaged, and delivered directly to program recipients in their homes.

SUMMARY:
The primary objective of this study is to evaluate the impact of provision of a child bed through the Beds for Kids program on objectively measured child sleep, and on daily child behavioral functioning and caregiver functioning over a 14-day period for preschool-aged children.

DETAILED DESCRIPTION:
Many lower-socioeconomic status (SES) children live in crowded homes and lack their own bed, which can contribute to insufficient and poor quality sleep and related poor child and family functioning. The Beds for Kids program provides beds and bedding to disadvantaged children in Philadelphia, and has been found to positively impact parent-reported child sleep in a previous pilot study. However, there is a need to determine the impact of the Beds for Kids program on objectively assessed child sleep, as well as on daily child behavior and caregiver functioning (mood and sleep). The primary objective of this study is to evaluate the impact of provision of a child bed through the Beds for Kids program on objectively measured child sleep, and on daily child behavioral functioning and caregiver functioning over a 14-day period for preschool-aged children. This is a randomized controlled trial (RCT). Caregiver-child dyads will be assigned to the intervention group, in which they receive a bed through the Beds for Kids program after a 7-day period, or to the waitlist control group, in which they receive a bed after a 14-day period. The primary study outcome is the difference between study conditions in actigraph-derived and caregiver-reported child sleep (bedtime, bedtime variability, sleep quality, night wakings, total sleep duration) for days 7 to 14 (bed vs control), as well as compared to baseline. Thus, this is a mixed between (bed vs waitlist) and within (days 1-7 vs days 8-14) group design.

ELIGIBILITY:
Inclusion Criteria:

* Males or females ages 2 to 5 years (24-71 months) and their male or female caregiver reporter (legal guardian)
* Eligible for the Beds for Kids program: (a) living without individual bedding (sleeping on the floor, on a sofa, or crowded into one bed with family members); (b) living in a household whose income is at or below 100 percent of the Federal Poverty Guideline.
* Parent/guardian is English-speaking.
* Caregiver is legal guardian and can complete informed consent.

Exclusion Criteria:

* Presence of a chronic medical (e.g., cancer, sickle cell disease) or neurodevelopmental (e.g., autism, Trisomy 21) that would impact sleep, including a pre-existing sleep disorder diagnosis (e.g., obstructive sleep apnea) in child.
* Child or caregiver use of prescription (e.g., clonidine) or over-the-counter medication (e.g., Benadryl; melatonin) that could impact the child's sleep or caregiver report of child's sleep.
* Caregivers/guardians or subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.

Ages: 24 Months to 71 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-02-03 (Actual); Study Completion 2020-02-03 (Actual)

PRIMARY OUTCOMES:
Child sleep duration | 14 day period
  Actigraph-derived child sleep duration in hours
Child sleep time variability | 14-day period
  Standard deviation of actigraph-derived child sleep time
Child sleep quality | 14-day period
  Caregiver-rated child sleep quality

SECONDARY OUTCOMES:
Child behavior problems (after 14-day period) | 14-day period
  Change in caregiver-rated daily child behavior problems
Caregiver emotional stress (after 14-day period) | 14-day period
  Change in caregiver-reported caregiver daily caregiver stress levels.
Child sleep duration at one-month follow-up | 6-7 weeks
  Change in caregiver-reported child sleep duration in hours from baseline (prior to actigraph/daily diary procedures) to one month post-bed delivery.
Child behavior problems at one-month follow-up | 6-7 weeks
  Change in caregiver-reported child behavior problems from baseline (prior to actigraph/daily diary procedures) to one month post-bed delivery: Child Behavior Checklist measure

CONTACTS AND LOCATIONS:
Overall Officials: Ariel A Williamson, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mindell JA, Sedmak R, Boyle JT, Butler R, Williamson AA. Sleep Well!: A Pilot Study of an Education Campaign to Improve Sleep of Socioeconomically Disadvantaged Children. J Clin Sleep Med. 2016 Dec 15;12(12):1593-1599. doi: 10.5664/jcsm.6338. PMID 27655459
- [Background] Bagley EJ, Kelly RJ, Buckhalt JA, El-Sheikh M. What keeps low-SES children from sleeping well: the role of presleep worries and sleep environment. Sleep Med. 2015 Apr;16(4):496-502. doi: 10.1016/j.sleep.2014.10.008. Epub 2014 Dec 16. PMID 25701537
- [Background] Hale L, Berger LM, LeBourgeois MK, Brooks-Gunn J. Social and demographic predictors of preschoolers' bedtime routines. J Dev Behav Pediatr. 2009 Oct;30(5):394-402. doi: 10.1097/DBP.0b013e3181ba0e64. PMID 19745760
- [Background] McLaughlin Crabtree V, Beal Korhonen J, Montgomery-Downs HE, Faye Jones V, O'Brien LM, Gozal D. Cultural influences on the bedtime behaviors of young children. Sleep Med. 2005 Jul;6(4):319-24. doi: 10.1016/j.sleep.2005.02.001. Epub 2005 Apr 1. PMID 15978515
- [Background] de Jong DM, Cremone A, Kurdziel LB, Desrochers P, LeBourgeois MK, Sayer A, Ertel K, Spencer RM. Maternal Depressive Symptoms and Household Income in Relation to Sleep in Early Childhood. J Pediatr Psychol. 2016 Oct;41(9):961-70. doi: 10.1093/jpepsy/jsw006. Epub 2016 Mar 19. PMID 26994853
- [Background] Meltzer LJ, Mindell JA. Relationship between child sleep disturbances and maternal sleep, mood, and parenting stress: a pilot study. J Fam Psychol. 2007 Mar;21(1):67-73. doi: 10.1037/0893-3200.21.1.67. PMID 17371111
- [Background] Van Dyk TR, Thompson RW, Nelson TD. Daily Bidirectional Relationships Between Sleep and Mental Health Symptoms in Youth With Emotional and Behavioral Problems. J Pediatr Psychol. 2016 Oct;41(9):983-92. doi: 10.1093/jpepsy/jsw040. Epub 2016 May 16. PMID 27189691
- [Background] Pena MM, Rifas-Shiman SL, Gillman MW, Redline S, Taveras EM. Racial/Ethnic and Socio-Contextual Correlates of Chronic Sleep Curtailment in Childhood. Sleep. 2016 Sep 1;39(9):1653-61. doi: 10.5665/sleep.6086. PMID 27306269
- [Background] Kushnir J, Sadeh A. Correspondence between reported and actigraphic sleep measures in preschool children: the role of a clinical context. J Clin Sleep Med. 2013 Nov 15;9(11):1147-51. doi: 10.5664/jcsm.3154. PMID 24235895
- [Background] Achenbach TM. The Achenbach System of Empirically Based Assessment (ASEBA): Development, Findings, Theory, and Applications. 2009; Burlington, VT: University of Vermont Research Center for Children, Youth, and Families.
- [Background] Radloff LS. The CES-D scale: a self-report depression scale for research in the general population. Appl Psychol Meas 1977;1:385-401.
- [Background] Sadeh A. The role and validity of actigraphy in sleep medicine: an update. Sleep Med Rev. 2011 Aug;15(4):259-67. doi: 10.1016/j.smrv.2010.10.001. Epub 2011 Jan 14. PMID 21237680
- [Result] Williamson AA, Min J, Fay K, Cicalese O, Meltzer LJ, Mindell JA. A multimethod evaluation of bed provision and sleep education for young children and their families living in poverty. J Clin Sleep Med. 2023 Sep 1;19(9):1583-1594. doi: 10.5664/jcsm.10614. PMID 37086055

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-21): https://cdn.clinicaltrials.gov/large-docs/44/NCT03392844/Prot_SAP_000.pdf